CLINICAL TRIAL: NCT00737594
Title: A Randomized, Placebo-controlled, Double-blinded Study of the Efficacy and Safety of Cobiprostone in Patients With Portal Hypertension
Brief Title: Efficacy and Safety of Cobiprostone in Patients With Portal Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to enroll a suitable number of qualified subjects.
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Sucampo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH0721
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2016-02

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — cobiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo TID (Placebo Comparator): Participants receive matching placebo capsules three times daily (TID)
  Interventions: Drug: Placebo
- 12 mcg TID (Experimental): Participants receive 12 mcg Cobiprostone TID
  Interventions: Drug: Cobiprostone
- 18 mcg TID (Experimental): Participants receive 18 mcg Cobiprostone TID
  Interventions: Drug: Cobiprostone

INTERVENTIONS:
Drug: Placebo — Matching placebo capsules for oral administration
  Other Names: Matching placebo
  Arms: Placebo TID
Drug: Cobiprostone — Cobiprostone capsules for oral administration
  Other Names: Experimental product
  Arms: 12 mcg TID; 18 mcg TID

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of cobiprostone (at two dose levels) as compared to placebo for lowering portal hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >= 18 years of age.
* Patient has clinical and/or pathological diagnosis of intra-hepatic portal hypertension.
* Patient has clinical diagnosis of cirrhosis.
* Patient has undergone variceal banding.

Exclusion Criteria:

* Patient has a Child-Pugh score >12.
* Patient has portal hypertension resulting from hepatic vein obstruction, portal vein occlusion, schistosomiasis, portal vein thrombosis, splenic vein thrombosis, or Budd-Chiari syndrome.
* Variceal banding procedure was performed within 1 month of the screening visit.
* Patient has active or recurrent variceal bleeding, or has had variceal bleeding within the 12 weeks prior to screening.
* Patient is unwilling to discontinue use of vasoactive drugs from the screening visit through the end of the study.
* Patient has hepatocellular carcinoma that is being medically treated or is advanced.
* Patient has impaired renal function (i.e., serum creatinine concentration >1.8 mg/dl)
* Patient has a history of liver transplant, or is expected to receive a liver transplant during the study period.
* Patient has undergone a gastrointestinal or abdominal surgical procedure within 90 days prior to the Screening Visit, or has had a bowel resection at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Investigator, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants were recruited, but the study terminated before data were collected
Groups:
- Placebo: Placebo: 0 mcg capsules three times daily (TID)
- 12 mcg TID: Cobiprostone 36 mcg
  Cobiprostone: 12 mcg cobiprostone (capsules) three times daily (TID)
- 18 mcg TID: Cobiprostone 54 mcg
  Cobiprostone: 18 mcg cobiprostone (capsules) three times daily (TID)
Period: Overall Study
Arm/Group | Placebo | 12 mcg TID | 18 mcg TID
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study terminated before data were collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 12 mcg TID | 18 mcg TID | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hepatic Venous Pressure Gradient (HVPG) After Four (4) Weeks of Treatment
Time Frame: 4 weeks
Population: Study terminated early, data were not collected.
Arm/Group | Placebo | 12 mcg TID | 18 mcg TID
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The trial terminated before data were collected
Description: The trial terminated before data were collected
Arm/Group | Placebo | 12 mcg TID | 18 mcg TID
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The trial terminated before data were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No